CLINICAL TRIAL: NCT07229313
Title: A Phase 1 Dose-Finding and Dose-Expansion Study of KIVU-107 in Participants With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of KIVU-107 in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kivu Bioscience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KIVU-107-01
Record Dates: First submitted 2025-09-16; First posted 2025-11-14 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Advance Solid Tumors
Keywords: PTK7; ADC; solid tumors; PTK-7 expression; metastatic; locally advanced; PTK7 expression; endometrial cancer; ovarian cancer; breast cancer; cervical cancer; GI/GEJ adenocarcinoma; esophageal squamous cell cancer; colorectal cancer; pancreatic cancer; non-small cell lung cancer; small cell lung cancer; head and neck squamous cell carcinoma; sarcoma; OvCa; NSCLC; SCLC; CRC; PDAC; HNSCC; TNBC; triple negative breast cancer; antibody drug conjugate
MeSH Terms: conditions — Neoplasm Metastasis; Endometrial Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms; Esophageal Squamous Cell Carcinoma; Colorectal Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Squamous Cell Carcinoma of Head and Neck; Sarcoma; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Finding (Experimental): Part A: KIVU-107 Dose Finding - Participants will be treated with KIVU-107 in multiple ascending cohorts.
  Interventions: Drug: KIVU-107
- Dose Expansion (Experimental): Part B: KIVU-107 Dose Expansion - Participants will be treated with the RDE from Part A.
  Interventions: Drug: KIVU-107

INTERVENTIONS:
Drug: KIVU-107 — KIVU-107 will be administered IV.

SUMMARY:
This is a 2-part, first-in-human, open-label study to determine the safety and tolerability of KIVU-107, a PTK7-directed antibody-drug conjugate, in participants with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
Part A: The primary objective of Part A of this study is to evaluate the safety and tolerability of KIVU-107 and to determine the maximum tolerated dose (MTD)/Recommended Dose for Expansion (RDE).

Part B: The primary objective of Part B of this study is to confirm the safety and tolerability of KIVU-107 at the RDE.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age
* No therapy of proven efficacy exists for the tumor
* Pathologically or histologically documented diagnosis of advanced / metastatic solid tumor malignancy that is resistant to standard therapy or for which no standard therapy is available.
* Adequate bone marrow, kidney, and liver function
* Measurable disease using RECIST v1.1
* ECOG 0 or 1
* Life expectancy ≥ 3 months

Exclusion Criteria:

* Prior treatment with any ADC with topoisomerase 1 inhibitor payload
* Any PTK7 - targeted therapy
* Uncontrolled cardiovascular disease
* Active Hepatitis B, Hepatitis C, or HIV infection
* History of interstitial lung disease
* Major surgery, radiation therapy, or systemic anti-cancer within 3 weeks of study treatment start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Part A (Dose Finding): To determine the Maximum Tolerated Dose (MTD) | Up to 18 months
  Number of participants with treatment emergent adverse events
Number of participants with treatment related adverse events as assessed by CTCAE version 5.0 | Up to 18 months
To evaluate safety and tolerability of KIVU-107 | Up to 30 months
  Number of participants with treatment related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) is percentage of participants with best response of complete response (CR) or partial response (PR) according to RECIST 1.1 | Up to 30 months
Duration of Response (DOR) | Up to 30 months
  Time from CR or PR to objective disease progression or death to any cause
To evaluate the immunogenicity as measured by change of anti-drug antibodies in participants treated with KIVU-107 | Up to 30 months
Maximum Serum concentration of KIVU-107 (Cmax) | 21 days
  PK assessment
Maximum serum concentration of KIVU-107 (Cmin) | 21 days
  PK assessment
Maximum Serum concentration of KIVU-107 at Steady State (Cmax, ss) | up to 168 days
  PK assessment
Minimum Serum Concentration of KIVU-107 at Steady State (Cmin, ss) | up to 168 days
  PK assessment
Time of Maximum Serum Concentration of KIVU-107 (Tmax) | up to 168 days
  PK assessment
Time of Minimum Serum Concentration of KIVU-107 (Tmin) | up to 168 days
  PK assessment
Time of Minimum Serum Concentration of KIVU-107 (Tmin, ss) | Up to 168 days
  PK assessment
Terminal Half-Life (t1/2) of Serum KIVU-107 | Up to 168 days
  PK assessment
Area under the Serum Concentration-Time curve from the time of dosing to the last measurable concentration (AUClast) for KIVU-107 | 21 days
  PK Assessment
Area under the Serum Concentration-Time curve from the time of dosing extrapolated to time infinity (AUCinf) for KIVU-107 | Up to 168 days
  PK Assessment
Clearance (CL) of KIVU-107 | Up to 168 days
  PK Assessment
Apparent volume of distribution during the terminal phase (Vz) of KIVU-107 | Up to 168 days
  PK Assessment
Accumulation ration (Rac) of KIVU-107 | Up to 168 days
  PK Assessment

OTHER OUTCOMES:
To evaluate biomarkers with potential to predict response and/or resistance to KIVU-107 characterize baseline levels and/ or changes in genomic, mRNA and/or protein biomarkers to determine any signatures correlated with response or resistance. | Up to 30 months
Progression Free Survival (PFS) is defined as the time from the first dose to either disease progression according to RECIST v. 1.1, or death due to any cause, whichever comes first. | Up to 30 months
Overall Survival (OS) | Up to 30 months
  Proportion of participants alive at 1 year from the start of treatment to death from any cause
Time to Response (TTR) | Up to 30 months
  Time from start of treatment to complete response or partial response
Disease Control Rate (DCR) | Up to 30 months
  Proportion of participants with CR, PR, or SD

CONTACTS AND LOCATIONS:
Overall Officials: Louie Naumovski, MD, PhD, Study Chair — Kivu Bioscience
Locations (3):
- Australia (3):
  - Kivu Trial Site, Sydney, New South Wales
  - Kivu Trial Site, Brisbane, Queensland
  - Kivu Trial Site, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research.